CLINICAL TRIAL: NCT05537987
Title: A Multicenter, Open-Label Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-723 in Patients With Advanced Solid Tumors
Brief Title: Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-723 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InnoCare Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00502
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ICP-723 (Experimental)
  Interventions: Drug: ICP-723

INTERVENTIONS:
Drug: ICP-723 — 3+3 dose escalation

SUMMARY:
During this study, dose escalation will be conducted in subjects with advanced solid tumors who have experienced treatment failure after clinical standard of care treatments or who currently have no effective treatment available to evaluate the safety, tolerability, and PK of ICP-723

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathologically confirmed locally advanced malignant solid tumors that are unresectable or metastatic and that are unresponsive to standard treatments or have relapsed; patients who have progressed under standard treatment including prior treatment with TRK or ROS1 inhibitors.
2. Male or female patients with age ≥18 years old and ≤80 years old.
3. Measurable lesion according to RECIST 1.1.
4. Adequate organ functions that meet protocol requirement criteria.
5. Patients with asymptomatic, stable primary central nervous system (CNS) tumors or CNS metastases (treated or untreated)
6. Participates voluntarily, signs informed consent, and follows the study treatment plan and scheduled visits.

Exclusion Criteria:

1. Other than the advanced malignant solid tumor under study, patients with another one or more active malignancies within the previous 5 years except for locally curable cancers that have been apparently cured
2. Received systemic anti-cancer therapy including chemotherapy (except for oral fluorouracil chemotherapy), radiation therapy, hormones, targeted drugs, or biological immunotherapy within 4 weeks or 5 half-lives
3. Major surgery (thoracotomy, laparotomy, etc.) within 4 weeks or minor surgery (superficial skin surgery, lymphadenectomy, hernia repair, etc.) within 2 weeks before the first dose of the study drug
4. Clinically significant gastrointestinal/neurological dysfunction that may affect drug intake, transport, or absorption.
5. Has evidence of uncontrolled heart disease
6. At the investigator's discretion, evidence of severe or uncontrolled systemic disease.
7. Other conditions considered by the investigator to be inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicity (DLT), adverse events (AEs), and serious adverse events (SAEs). Frequency of dose interruptions, reductions and intensity | through study completion, an average of 1.5 years.

SECONDARY OUTCOMES:
Objective response rate (ORR) determined using RECIST 1.1 criteria. | Through study completion, an average of 4 years
Disease control rate (DCR) determined using RECIST 1.1 criteria. | Through study completion, an average of 4 years
Peak concentration (Cmax) | Through study completion, an average of 4 years
Time to reach peak concentration (Tmax) | Through study completion, an average of 4 years
Half-life (t1/2) | Through study completion, an average of 4 years
Area under the plasma concentration-time curve (AUC0-∞ and AUC0-t) | Through study completion, an average of 4 years
Apparent clearance (CL/F) | Through study completion, an average of 4 years
Apparent volume of distribution (Vz/F), | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Principal Investigator — University of Kansas Medical / Cancer Centers
Locations (3):
- United States (3):
  - University of Kansas Medical / Cancer Centers, Kansas City, Kansas
  - NYU-Langone Medical Center, New York, New York
  - Northwest Medical Specialties, Tacoma, Washington